CLINICAL TRIAL: NCT02369055
Title: Relationship Between Quality of Life and Rehabilitation Pathway One Year Post Stroke in Northern Norway and Denmark. A Mixed Method Study.
Brief Title: Quality of Life and Rehabilitation Pathway in Northern Norway and Denmark.
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: SFP1174-14
Record Dates: First submitted 2015-01-13; First posted 2015-02-23 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Quality of Life
Keywords: Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke survivors in North Norway: Patients with ischemic or heamorrhagic stroke admitted to stroke units in UNN Tromso, Narvik or Harstad (Norway), and living in the defined geographic area of these 3 hospitals.
- Stroke survivors in Denmark: Patients with ischemic og heamorrhagic stroke admitted to a stroke unit in Aarhus University Hospital and living in the municipalities of Randars or Favrskov in Central Denmark Region

SUMMARY:
The aim of this study is to analyze and describe rehabilitation pathways of stroke patients in a region of North Norway and Central Denmark Region in relation to how patients perceive quality of life, health and functioning one year post stroke.

The study will consist of 1) Translate, cross-cultural adapt and validate a stroke-specific health-related questionnaire 2) Describe the level of quality of life and rehabilitation pathway in the two countries 3) In-depth interviews of a smaller group of patients for a more complex understanding

The study is part of a larger prospective observational multicenter-study of two patient cohorts with stroke.

DETAILED DESCRIPTION:
Anticipated: 500 patients from Norway and 500 patients from Denmark are included in the national stroke-register datasets, and 250 patients from each country in the questionnaire-based datasets.

The questionnaire includes demographic data, the Stroke-Specific Quality of Life (SS-QOL) scale, Hospital Anxiety and Depression Scale (HADS), The EuroQol Quality of Life scale (EQ-5D), the EuroQol Visual Analogue Scale (EQ-VAS), the Quality of Life After Brain Injury, Overall Scale QOLIBRI-OS, modified Rankin Scale (mRS), and additional questions about satisfaction on treatment and rehabilitation.

5-6 patients from each country will be selected for semi-structured interviews with both priori questions and exploratory questions.

The mixing of methods will balance the goals of generality and complex understanding in how patients describe their quality of life and rehabilitation-chain.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the hospitals; UNN Tromso,Harstad, Narvik (Norway) and Aarhus (Denmark).

Exclusion Criteria:

Unverified stroke and residence outside of the studyregion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stroke
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life | one year
  The Stroke-Specific Quality of Life (SS-QOL) scale

CONTACTS AND LOCATIONS:
Overall Officials: Audny Anke, PhD, Study Chair — Division of Rehabilitation Services, University Hospital of North
Locations (1):
- Universitetet i Tromsø, Norges Arktiske Universitet, Det helsevitenskapelige fakultet, Institutt for helse og omsorgsfag, Tromsø, Norway